CLINICAL TRIAL: NCT00017524
Title: A Phase I Dose-Escalation Study of AG2037 Administered Once Weekly for Three Weeks to Patients With Advanced Cancer
Brief Title: AG2037 in Treating Patients With Advanced, Metastatic, or Recurrent Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068699; UAB-0052; AG-2037-003-A2; UAB-F001227008; NCI-G01-1954
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2012-11

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — pelitrexol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: pelitrexol

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of AG2037 in treating patients who have advanced, metastatic, or recurrent solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and dose-limiting toxic effects of AG2037 in patients with advanced, metastatic, or recurrent solid tumor.
* Determine the safety and tolerance of this drug in these patients.
* Assess the pharmacokinetics of this drug in these patients.
* Document any antitumor effects of this drug in these patients.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive AG2037 IV weekly on weeks 1-3. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of AG2037 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity.

Patients are followed weekly for 4 weeks.

PROJECTED ACCRUAL: A total of 18-60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed solid tumor

  * Advanced, metastatic, or recurrent disease
  * No curative therapy exists
* Measurable or evaluable disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* WHO 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL

Hepatic:

* Bilirubin no greater than 1.5 mg/dL (unless due to Gilbert's syndrome)
* SGOT OR SGPT no greater than 2 times upper limit of normal (ULN) (5 times ULN if liver metastases present)

Renal:

* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min

Other:

* No unstable or severe concurrent medical condition that would preclude study participation
* No sociological or familial condition that would preclude study compliance
* No psychological or addictive disorder that would preclude study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosourea or mitomycin) and recovered

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered
* No prior radiotherapy to more than 40% of bone marrow

Surgery:

* Not specified

Other:

* At least 2 weeks since prior blood transfusions
* At least 4 weeks since prior investigational agent and recovered
* No prior glycinamide ribonucleotide formyltransferase (GARFT) inhibitor
* No concurrent extradietary folate supplements
* No concurrent allopurinol
* No other concurrent anticancer or investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2001-03; Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Robert, MD, FACP, Study Chair — University of Alabama at Birmingham
Locations (3):
- United States (3):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida